CLINICAL TRIAL: NCT05801328
Title: Comparison Between Occlusal Versus Apical Bent Wires in Patients on Erich Arch Bar: A Prospective Split-mouth Randomized Clinical Trial
Brief Title: Comparison Between Occlusal Versus Apical Bent Wires in Patients on Erich Arch Bar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Ng Kar Tsyeng, Principal investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USM/JEPeM/22110704
Record Dates: First submitted 2023-03-12; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Maxillofacial Injuries
MeSH Terms: conditions — Maxillofacial Injuries

STUDY DESIGN:
Intervention Model Description: this is a split mouth study. Participants teeth will be divided into left or right side and randomised into either control or intervention side.
Who Masked: Participant
Masking Description: Participants are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occlusal ending of wires (Experimental): The wires will be bent occlusally for the interventional side
  Interventions: Device: Ending of the wires on Erich arch bar in the occlusal direction
- Apical ending of wires (No Intervention): The wires will be bent apically for the control side.

INTERVENTIONS:
Device: Ending of the wires on Erich arch bar in the occlusal direction — The wires of the Erich arch bar will be placed on the occlusal direction
  Arms: Occlusal ending of wires

SUMMARY:
Patients with jaw fractures requires placement of Erich arch bar for immobilization of the fractured jaw. However, the usage of Erich arch bar is associated with an increased in the incidence of mucosal trauma and plaque accumulation. Conventionally, the ends of the wires has always been placed apical to the teeth.

This study aims to determine if a change in the placement of the wire by directing it to the occlusal direction will reduce the incidence of mucosal trauma, plaque accumulation and if the stability of the Erich arch bar will be affected by this intervention.

The patients' teeth will be divided into left and right side and randomized into control side (wires end apically) and interventional side (wires end occlusally)

ELIGIBILITY:
Inclusion Criteria:

* 18 years - 60 years old.
* Full Glasgow coma scale.
* Facial fractures requiring Erich arch bar for 4 weeks duration
* No functional deficit that will prevent tooth brushing.

Exclusion Criteria:

* All pathologic fractures due to cysts, tumors, and cancers
* Medical conditions that contraindicate the usage of arch bars (Epilepsy, Asthmatics)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Are there any differences between occlusally and apically bent groups in terms of mucosal trauma? | Assessed on the second week
  Any mucosal injuries (Indentations, Entrapment, ulcerations) during follow up will be recorded as scored as '1'.
Are there any differences between occlusally and apically bent groups in terms of mucosal trauma? | Assessed on the fourth week
  Any mucosal injuries (Indentations, Entrapment, ulcerations) during follow up will be recorded as scored as '1'.

SECONDARY OUTCOMES:
Are there any differences between occlusally and apically bent groups in terms of Turesky-Gilmore-Glickman plaque score? | Assessed on the fourth week.
  Assessment of the plaque score using Turesky-Gilmore-Glickman plaque score.
  There are 6 scores for this plaque index, ranging from score '0' to '5'. Score '0' means that no plaque is seen, '1' when separate flecks of plaque at the cervical margin of the tooth, '2' when a thin continuous band of plaque at the cervical margin of the tooth, '3' when a band of plaque thicker than 1mm but less than 1/3rd of the tooth surface. '4' when plaque covers at least 1/3rd but less than 2/3rd of the crown and '5' when plaque is covering 2/3rd or more of the crown of the tooth. The teeth involved in the scoring in this study are buccal surfaces of the 1st molars, premolars, canines and incisors. Since the lingual/palatal surfaces are not accessible as the teeth are wired up, it will not be assessed
  Score '0' is the best while score of '5' is the worst.
  This assessment is done on the fourth week after removal of the arch bar and staining of the teeth with a disclosing solution.
Are there any differences between occlusally and apically bent groups in terms of stability of the arch bar? | Assessed on the second week
  The operator will assess all circumferential wires on the second week. Any loose wires will be scored as '1' and '0' if the wires are firm.
  The loose wires will be retightened.
Are there any differences between occlusally and apically bent groups in terms of stability of the arch bar? | Assessed on the fourth week
  The operator will assess all circumferential wires on the fourth week. Any loose wires will be scored as '1' and '0' if the wires are firm.
  The loose wires will be retightened.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adeyemo WL, Ladeinde AL, Ogunlewe MO, James O. Trends and characteristics of oral and maxillofacial injuries in Nigeria: a review of the literature. Head Face Med. 2005 Oct 4;1:7. doi: 10.1186/1746-160X-1-7. PMID 16270942
- [Background] Qureshi AA, Reddy UK, Warad NM, Badal S, Jamadar AA, Qurishi N. Intermaxillary fixation screws versus Erich arch bars in mandibular fractures: A comparative study and review of literature. Ann Maxillofac Surg. 2016 Jan-Jun;6(1):25-30. doi: 10.4103/2231-0746.186129. PMID 27563602
- [Background] Bali R, Sharma P, Garg A. Incidence and patterns of needlestick injuries during intermaxillary fixation. Br J Oral Maxillofac Surg. 2011 Apr;49(3):221-4. doi: 10.1016/j.bjoms.2010.04.010. Epub 2010 May 21. PMID 20488595
- [Background] de Queiroz SB. Modification of arch bars used for intermaxillary fixation in oral and maxillofacial surgery. Int J Oral Maxillofac Surg. 2013 Apr;42(4):481-2. doi: 10.1016/j.ijom.2012.11.003. Epub 2012 Dec 12. PMID 23245627
- [Background] Farber SJ, Snyder-Warwick AK, Skolnick GB, Woo AS, Patel KB. Maxillomandibular Fixation by Plastic Surgeons: Cost Analysis and Utilization of Resources. Ann Plast Surg. 2016 Sep;77(3):305-7. doi: 10.1097/SAP.0000000000000592. PMID 26207551
- [Background] Fasoulas A, Pavlidou E, Petridis D, Mantzorou M, Seroglou K, Giaginis C. Detection of dental plaque with disclosing agents in the context of preventive oral hygiene training programs. Heliyon. 2019 Jul 10;5(7):e02064. doi: 10.1016/j.heliyon.2019.e02064. eCollection 2019 Jul. PMID 31334380
- [Background] Fernandes IA, Lopes ABS, Fonseca PG, da Silva Torres A, Rodrigues AB, Galvao EL, Falci SGM. Comparison between Erich arch bars and intermaxillary screws in maxillofacial fractures involving the dental occlusion: a meta-analysis. Int J Oral Maxillofac Surg. 2021 Jan;50(1):83-95. doi: 10.1016/j.ijom.2020.07.022. Epub 2020 Aug 12. PMID 32798159
- [Background] Garra G, Singer AJ, Taira BR, Chohan J, Cardoz H, Chisena E, Thode HC Jr. Validation of the Wong-Baker FACES Pain Rating Scale in pediatric emergency department patients. Acad Emerg Med. 2010 Jan;17(1):50-4. doi: 10.1111/j.1553-2712.2009.00620.x. Epub 2009 Dec 9. PMID 20003121
- [Background] Gilardino MS, Chen E, Bartlett SP. Choice of internal rigid fixation materials in the treatment of facial fractures. Craniomaxillofac Trauma Reconstr. 2009 Mar;2(1):49-60. doi: 10.1055/s-0029-1202591. No abstract available. PMID 22110797
- [Background] Haggard P, de Boer L. Oral somatosensory awareness. Neurosci Biobehav Rev. 2014 Nov;47:469-84. doi: 10.1016/j.neubiorev.2014.09.015. Epub 2014 Oct 2. PMID 25284337
- [Background] Hamid ST, Bede SY. The Use of Screw Retained Hybrid Arch Bar for Maxillomandibular Fixation in the Treatment of Mandibular Fractures: A Comparative Study. Ann Maxillofac Surg. 2021 Jul-Dec;11(2):247-252. doi: 10.4103/ams.ams_35_21. Epub 2022 Feb 1. PMID 35265493
- [Background] Jain A, Taneja S, Rai A. What is a better modality of maxillomandibular fixation: bone-supported arch bars or Erich arch bars? A systematic review and meta-analysis. Br J Oral Maxillofac Surg. 2021 Oct;59(8):858-866. doi: 10.1016/j.bjoms.2021.01.004. Epub 2021 Jan 18. PMID 34315565
- [Background] Kirk D, Whitney J, Shafer D, Song L. Tight Placement of Erich Arch Bar While Avoiding Wire Fatigue Failure. J Oral Maxillofac Surg. 2016 Mar;74(3):562-8. doi: 10.1016/j.joms.2015.10.008. Epub 2015 Oct 19. PMID 26546844
- [Background] Koshy JC, Feldman EM, Chike-Obi CJ, Bullocks JM. Pearls of mandibular trauma management. Semin Plast Surg. 2010 Nov;24(4):357-74. doi: 10.1055/s-0030-1269765. PMID 22550460
- [Background] Loe H. Oral hygiene in the prevention of caries and periodontal disease. Int Dent J. 2000 Jun;50(3):129-39. doi: 10.1111/j.1875-595x.2000.tb00553.x. PMID 10967765
- [Background] Tracy K, Gutta R. Are embrasure wires better than arch bars for intermaxillary fixation? J Oral Maxillofac Surg. 2015 Jan;73(1):117-22. doi: 10.1016/j.joms.2014.08.020. Epub 2014 Aug 27. PMID 25511963
- [Background] Uhthoff HK, Poitras P, Backman DS. Internal plate fixation of fractures: short history and recent developments. J Orthop Sci. 2006 Mar;11(2):118-26. doi: 10.1007/s00776-005-0984-7. PMID 16568382
- [Background] Vadepally AK, Sinha R. Is it better to bend wires occlusally or apically during placement of arch bars for intermaxillary fixation? Br J Oral Maxillofac Surg. 2018 Jan;56(1):67-69. doi: 10.1016/j.bjoms.2017.11.006. Epub 2017 Dec 6. PMID 29198481
- [Background] van den Bergh B, Blankestijn J, van der Ploeg T, Tuinzing DB, Forouzanfar T. Conservative treatment of a mandibular condyle fracture: Comparing intermaxillary fixation with screws or arch bar. A randomised clinical trial. J Craniomaxillofac Surg. 2015 Jun;43(5):671-6. doi: 10.1016/j.jcms.2015.03.010. Epub 2015 Mar 27. PMID 25911121
- [Background] Kaura S, Kaur P, Bahl R, Bansal S, Sangha P. Retrospective Study of Facial Fractures. Ann Maxillofac Surg. 2018 Jan-Jun;8(1):78-82. doi: 10.4103/ams.ams_73_17. PMID 29963429
- [Background] Saperi BS, Ramli R, Ahmed Z, Muhd Nur A, Ibrahim MI, Rashdi MF, Nordin R, Rahman NA, Yusoff A, Nazimi AJ, Abdul Rahman R, Abdul Razak N, Mohamed N. Cost analysis of facial injury treatment in two university hospitals in Malaysia: a prospective study. Clinicoecon Outcomes Res. 2017 Feb 7;9:107-113. doi: 10.2147/CEOR.S119910. eCollection 2017. PMID 28223831
- [Background] Rothe TM, Kumar P, Shah N, Shah R, Mahajan A, Kumar A. Comparative Evaluation of Efficacy of Conventional Arch Bar, Intermaxillary Fixation Screws, and Modified Arch Bar for Intermaxillary Fixation. J Maxillofac Oral Surg. 2019 Sep;18(3):412-418. doi: 10.1007/s12663-018-1110-7. Epub 2018 Apr 19. PMID 31371884
- [Background] Rai A, Jain A, Datarkar A, Bhawalkar A. Use of oral screen for preventing soft tissue injuries associated with use of arch bars: a prospective randomized clinical study. Oral Maxillofac Surg. 2019 Sep;23(3):291-295. doi: 10.1007/s10006-019-00780-3. Epub 2019 May 16. PMID 31093796
- [Background] Pedemonte C, Valenzuela K, Gonzalez LE, Vargas I, Noguera A. Types of Intermaxillary Fixation and Their Interaction With Palatine Fracture Reduction. J Oral Maxillofac Surg. 2019 Oct;77(10):2083.e1-2083.e8. doi: 10.1016/j.joms.2019.06.006. Epub 2019 Jun 21. PMID 31310733
- See also: The Acute Management of Facial Fractures — https://www.infona.pl/resource/bwmeta1.element.springer-doi-10_1007-S40719-016-0040-4